CLINICAL TRIAL: NCT04737746
Title: Caregiver Burden and Correlation With Clinical Outcome in Spinal Cord
Brief Title: Caregiver Burden and Correlation With Clinical Outcome in Spinal Cord Stimulation for Chronic Neuropathic Pain
Acronym: CAREstim
Status: Completed | Type: Observational
Sponsor: AZ Delta (Other)
Responsible Party: Principal Investigator, Dimitri Vanhauwaert, neurosurgeon, AZ Delta
Other Study IDs: B1172020000048; CME AZ Delta (Other: Studie 20130)
Record Dates: First submitted 2021-01-26; First posted 2021-02-04 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Pain, Chronic; Pain, Neuropathic; Failed Back Surgery Syndrome
MeSH Terms: conditions — Chronic Pain; Neuralgia; Failed Back Surgery Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 13 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Prospective multicentric observational trial on caregiver burden, caregiver satisfaction and clinical outcome in spinal cord stimulation for chronic neuropathic pain.

DETAILED DESCRIPTION:
Spinal cord stimulation is an effective therapy for chronic neuropathic pain. After careful selection, the satisfaction for the patient is often considerable. The investigators want to investigate the caregiver burden for relatives of patients who are treated with spinal cord stimulation. This will be evaluated by appropriate scores at baseline, during neurostimulator trial and 3,6 and 12 months after implantation. At the same time the patient satisfaction and pain reduction will also be evaluated independently.

In this prospective cohort different parameters will be assessed at baseline, trial, 3, 6 and 12 months follow-up for the patient and their caregiver.

For the patient this will include Numeric Rating scale (NRS) for leg and back pain, Oswestry Disability Index (ODI), EuroQuality of Life-5 Dimensions score (EQ5D), opiate use and Relation Quality Index (RQI).

For the caregiver the Zarit Burden Index (ZBI), Relation Quality Index (RQI) and Modified Caregiver Strain Index (MCSI).

With regard to the research questions, subgroup analysis will be performed regarding to age, sex, education, neurostimulation pattern, surgical vs percutaneous lead placement, working status of both patient and caregiver and caregiver relation characteristics.

ELIGIBILITY:
Inclusion Criteria:

* Patients Age > 18 years
* Patients with an identified spousal or offspring caregiver
* Patients receiving neurostimulator for the first time
* Patient complies to reimbursement criteria for spinal cord stimulation in Belgium

Exclusion Criteria:

* Non-spinal cord type of neuromodulation (DRG, occipital, peripheral nerve, )
* Revision cases, previous neuromodulation
* Patients unable to consent for this study
* Patients without identified spousal or offspring caregiver

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who are considered to be treated with spinal cord stimulation in AZ Delta hospital and Jan Yperman hospital between 1/1/2021 and 31/12/2021 are potentially eligible for inclusion. The inclusion is not limited to a specific device and all different types of routinely used spinal cord stimulation systems and neurostimulation modalities are included: percutaneous of surgical lead placement in both thoracic or cervical location. All patients follow the standard flow for screening and reimbursement (neuro pain platform and MAO)
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2021-01-18 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Zarit Burden index | baseline to 12 months
  Zarit Burden index measures the burden of a caregiver in 12 questions
relation quality index caregiver | baseline to 12 months
caregiver strain index | baseline to 12 months

SECONDARY OUTCOMES:
NRS pain leg and back | baseline to 12 months
  numeric rating scale
Oswestry Disability Index | baseline to 12 months
EuroQol five dimensions EQ-5D | baseline to 12 months
relation quality index patient | baseline to 12 months
analgetics dose | baseline to 12 months
  analgetics ( paracetamol, opiates, opioids, non steroidal anti inflammatory and anti neuropathic pain medication

CONTACTS AND LOCATIONS:
Locations (2):
- Belgium (2):
  - Jan Ypermanziekenhuis, Ieper
  - AZ Delta, Roeselare

IPD SHARING:
Plan to Share IPD: No